CLINICAL TRIAL: NCT04011254
Title: Examining Salt Appetite in Haemodialysis Patients Using Functional Magnetic Resonance Imaging
Brief Title: Haemodialysis fMRI Salt Appetite Study
Acronym: HeMSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Yale University (Other); Forschungszentrum Juelich (Other)
Responsible Party: Sponsor
Other Study IDs: 19HH5153
Record Dates: First submitted 2019-06-25; First posted 2019-07-08 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Dialysis; Excess Interdialytic Weight Gain
Keywords: salt taste preference; salt taste sensitivity; functional Magnetic Resonance Imaging; Dialysis; Salt taste; salt intake
MeSH Terms: interventions — Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Control: Healthy control
- Haemodialysis %IDWG >4%: Patient on regular haemodialysis with average IDWG >4%
  Interventions: Procedure: haemodialysis
- Haemodialysis %IDWG <4%: Patient on regular haemodialysis with average IDWG <4%
  Interventions: Procedure: haemodialysis

INTERVENTIONS:
Procedure: haemodialysis — Routine haemodialysis session
  Groups: Haemodialysis %IDWG <4%; Haemodialysis %IDWG >4%

SUMMARY:
1. Assessing how the rapid removal of salt and water by haemodialysis alters regional brain activity (by measurement of the brain blood oxygen level-dependent (BOLD) signal using functional MRI) during tasting of soup of differing salt concentrations.
2. Identify differences in the brain response to salt taste pre- and post-haemodialysis between haemodialysis patients who are either able or unable to control between dialysis weight gain

DETAILED DESCRIPTION:
HeMSA Study Phase 2 Up to 20 male, haemodialysis patient who have average %IDWG >4% will be recruited with the target, to proceed to scanning, of 14 patients. Following consent the patients will complete questionnaires (including Salt intake questionnaire - DSQ (Gkza and Davenport, 2017), Edinburgh handedness questionnaire (Oldfield, 1971), MRI checklist) and undergo salt taste preference and threshold testing during a 1 hour session prior to dialysis. The purpose of this visit is to establish the tasteless solution and 2 soup salt concentrations to be used in the salt taste fMRI paradigm, obtain baseline data regarding estimate of salt intake and ensure MRI is safe for this patient.

Patients will then attend 2 MRI scanning visits at the Hammersmith Hospital Imperial Campus, one the morning immediately before haemodialysis and one the morning after haemodialysis. Prior to the MRI session, at the Imperial College Clinical Research Facility, the patient will undergo various clinical assessments and have venous blood samples taken. The MRI will be undertaken at the Imperial College Clinical Imaging Facility using a Siemens 3T Verio scanner. During the scan subjects will taste, via a taste delivery system, aliquots of tasteless solution, sucralose, and 2 soup with different concentrations of salt. Solutions will be delivered in a block design.

HeMSA Study Phase 3 3 groups (healthy controls, haemodialysis (HD) patients with %IDWG <4%, haemodialysis patients with %IDWG >4% - patients froms phase 2 will contribute to the latter group) Protocol will follow that for HeMSA Phase 2. Healthy controls will also have 2 study visits at a similar period apart to the HD participants.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Male
* Aged 18-65 years
* Non-smoker (ex-smokers allowed)
* Right handed (able to use a right handed response button)
* Able to tolerate 1 hour MRI scanning session

For haemodialysis patients:

* Established on haemodialysis for more than 6 months
* Urine output <200ml/24 hours
* Average (over the past month) interdialytic weight gain:

  1. Main phase 2: >4 %IDWG
  2. Main phase 3: <4 or >4 %IDWG

Exclusion Criteria:

* Type 1 or type 2 diabetes mellitus
* Current smoker
* Uncontrolled depression (change in use of anti-depressants in last 3 months, or BDI-II score >28/63)
* Neurological disorder (Parkinson's disease, serious cerebrovascular disease, epilepsy, moderate-severe traumatic brain injury, dementia)
* Previous bariatric surgery
* Inflammatory state (CRP >20 on routine dialysis blood tests)
* Acute infective illness
* Significant current or past medical or psychiatric history, or use of medications, that, in the opinion of the Investigators, contraindicates their participation, due to influence on outcome measures.
* Patients lacking capacity or unable to consent and non-English language speakers
* Contra-indication to MRI imaging e.g. metal insert, pacemaker
* Claustrophobia
* Patients currently participating in an active CTIMP trial, or within 4 half-lives of last administration of CTIMP product
* Serious mental illness (e.g. bipolar disorder, schizophrenia)
* Current alcohol or drug dependence

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Haemodialysis patients under the care of Imperial College NHS Healthcare Trust and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-02-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in regional brain BOLD signal during tasting of soup of differing salt concentrations (vs. artificial saliva) pre dialysis session verse post dialysis session | 1 week (maximal time between pre and post dialysis scan)
  Regional brain BOLD signal during tasting of soup of differing salt concentrations (vs. artificial saliva) ROI including insula, amygdala, ventral tegmental area, pre frontal cortex,

SECONDARY OUTCOMES:
Change in ratings of salt liking and intensity across different salt concentrations of soup | 1 week (maximal time between pre and post dialysis scan)
  Ratings of liking, via Labelled Hedonic Scale (LHS) (-100=Most disliked sensation imaginable, 0=neural, 100=Most liked sensation imaginable), of salted soup of 2 concentrations pre dialysis session verse post dialysis session
Change in ratings of sweet liking and intensity pre dialysis session verse post dialysis session | 1 week (maximal time between pre and post dialysis scan)
  Ratings of liking and intensity, via Labelled Hedonic Scale (LHS) (-100=Most disliked sensation imaginable, 0=neural, 100=Most liked sensation imaginable), of sucralose solution
Ratings of sour liking and intensity | 1 week (maximal time between pre and post dialysis scan)
  Rating of liking and intensity, via Labelled Hedonic Scale (LHS) (-100=Most disliked sensation imaginable, 0=neural, 100=Most liked sensation imaginable) of citrate pre dialysis session verse post dialysis session
Salt threshold testing | 1 week (maximal time between pre and post dialysis scan)
  The lowest concentration of saline solution detected by taste. pre dialysis session verse post dialysis session
Arterial spin labelling | 1 week (maximal time between pre and post dialysis scan)
  arterial spin labelling measurement of regional cerebral blood flow at rest pre dialysis session verse post dialysis session
cerebral vascular reactivity pre dialysis session verse post dialysis session | 1 week (maximal time between pre and post dialysis scan)
  BOLD signal changes during breath hold to assess BOLD signal reactivity to increased CO2 concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor C Sandhu, MBBS, Principal Investigator — Imperial College London; Tony Goldstone, MRCP PhD, Study Director — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No